CLINICAL TRIAL: NCT01759862
Title: Perioperative Aminophylline to Improve High Risk Renal Graft Outcome- a Double Blinded, Placebo Controlled, Randomized Clinical Trial
Brief Title: Perioperative Aminophylline to Improve Early Kidney Function After a Kidney Transplant
Acronym: RTphylline
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Orly Haskin, Pediatric Nephrology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24280
Record Dates: First submitted 2012-12-30; First posted 2013-01-03 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Function of Renal Transplant
Keywords: kidney transplant; Aminophylline; pediatric
MeSH Terms: interventions — Aminophylline; Theophylline; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aminophylline (Experimental): Patients will receive aminophylline loading dose 5mg/kg prior to transplant and will continue to receive aminophylline 1.8mg/kg Q6h for a total of 20 doses.
  Theophylline drug levels will be monitored daily for 4 days.
  Interventions: Drug: Aminophylline; Other: Theophylline drug levels
- Control (Placebo Comparator): Patients will receive placebo infusion of normal saline, pre-transplant, followed by normal saline infusions matched by volume and frequency to treatment arm for a total of 20 doses.
  Drug levels will be monitored daily for 4 days.
  Interventions: Other: Theophylline drug levels; Drug: Placebo

INTERVENTIONS:
Drug: Aminophylline — Aminophylline loading dose 5mg/kg prior to transplant and will continue to receive aminophylline 1.8mg/kg Q6h for a total of 20 doses.
  Other Names: Theophylline
  Arms: Aminophylline
Other: Theophylline drug levels — Theophylline drug levels will be monitored every morning from all patients for the first 4 days post- transplant.
Drug: Placebo — Patients will receive placebo infusion of normal saline, pre-transplant, followed by normal saline infusions matched by volume and frequency to treatment arm for a total of 20 doses.
  Other Names: Normal saline
  Arms: Control

SUMMARY:
The aim of this study is to evaluate whether peri-transplant administration of a drug named aminophylline to children undergoing a kidney transplant from deceased donors improves early graft function and also projects on long term graft function.

DETAILED DESCRIPTION:
This is a Double-blinded, placebo-controlled, randomized, clinical trial to evaluate whether administration of aminophylline starting pretransplant until post-transplant day 5 improves early kidney function and projects also on long term graft function.

Study Arms and intervention: On admit to the hospital prior to transplant, patients will be randomized into treatment or control arms. The randomization will be based on age groups 1-5y, 5-12y and 12-18y Treatment arm: Patients will receive aminophylline loading dose 5mg/kg prior to transplant and will continue to receive aminophylline 1.8mg/kg Q6h for a total of 20 doses.

Control arm: Patients will receive placebo infusion of normal saline, pre-transplant, followed by normal saline infusions matched by volume and frequency to treatment arm for a total of 20doses.

The only difference between the two arms will be the study intervention. Other than that all patients will receive the same standard of care for patients undergoing a kidney transplant.

Theophylline drug levels will be monitored every morning from all patients for the first 4 days post- transplant. Theophylline levels will be reported independently by the laboratory in a faxed research report directly to the pharmacist who will perform dose adjustments, according to the following table.

Theophylline Level (mcg/ml) Dose Adjustment <2 Increase subsequent doses by 50% 2-2.9 Increase subsequent doses by 33% 3-3.9 Increase subsequent doses by 25% 4-4.9 Increase subsequent doses by 15% 5-7 (goal) Target Level; No dose adjustment 7.1-8.4 Decrease subsequent doses by 10% 8.5-9.9 Decrease subsequent doses by 15% 10-12.4 Decrease subsequent doses by 25% 12.5-14.9 Decrease subsequent doses by 50% 15-19.9 Decrease subsequent doses by 67% >19.9 Discontinue all aminophylline doses. Contact Medical Monitor

All involved personnel will be blinded to the patient's allocation and to the drug level results.

The investigators will also collect a urine sample for NGAL (Neutrophil gelatinase-associated lipocalin)levels from all patients at 12 hours post-transplant.

Primary outcome will be calculated Glomerular Filtration Rate(GFR) on postoperative day 5. The investigators will determine whether patients in the aminophylline group had improved GFR compared to control group.

The investigators will also determine whether patients who received aminophylline had lower urinary NGAL levels compared to control group indicating a lesser degree of kidney injury. Urinary NGAL (Neutrophil gelatinase-associated lipocalin) is a biomarker of kidney injury. Elevated urinary NGAL levels post-transplant were found to be predictive of delayed graft function and the need for dialysis post-transplant.

At the investigators' center all patients undergo routine kidney protocol biopsies at 6 months post- transplant. After the slides are read by the pathologist the investigators will use the same tissue blocks to quantify the amount of fibrosis using computerized image analysis of Sirius Red-stained biopsies. The amount of fibrosis seen on 6 months protocol biopsies was proven to be correlated with expected graft survival.

An independent medical monitor will be assigned to manage toxic theophylline levels >20mcg/mL. The laboratory will report directly to the medical monitor, who will discontinue aminophylline and remove the patient from the study.

The trial will be also be monitored with a Data Safety Monitoring Board (DSMB) unrelated to the study. The DSMB will meet after enrollment of 20 patients to assess for drug safety and monitor for adverse events of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric kidney transplant recipients less than 21 years of age
2. Patients undergoing deceased donor (DD) kidney transplants

Exclusion Criteria:

1. Known history of non-sinus tachycardia
2. Multiple organ transplants recipients
3. Severe liver dysfunction
4. graft was placed on pump after harvesting

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2012-11; Primary Completion 2017-01-05 (Actual); Study Completion 2017-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul C Grimm, MD, Study Director — Medical director, Pediatric Kidney Transplant Program Department of Pediatric Nephrology , Lucile Packard Children's hospital
Locations (1):
- Lucile Packard Children's Hospital at Stanford, Stanford, California, United States

REFERENCES:
- [Background] Grenz A, Baier D, Petroktistis F, Wehrmann M, Kohle C, Schenk M, Sessler M, Gleiter CH, Fandrich F, Osswald H. Theophylline improves early allograft function in rat kidney transplantation. J Pharmacol Exp Ther. 2006 May;317(2):473-9. doi: 10.1124/jpet.105.096917. Epub 2006 Jan 12. PMID 16410406
- [Background] Bhat MA, Shah ZA, Makhdoomi MS, Mufti MH. Theophylline for renal function in term neonates with perinatal asphyxia: a randomized, placebo-controlled trial. J Pediatr. 2006 Aug;149(2):180-4. doi: 10.1016/j.jpeds.2006.03.053. PMID 16887430
- [Background] Jenik AG, Ceriani Cernadas JM, Gorenstein A, Ramirez JA, Vain N, Armadans M, Ferraris JR. A randomized, double-blind, placebo-controlled trial of the effects of prophylactic theophylline on renal function in term neonates with perinatal asphyxia. Pediatrics. 2000 Apr;105(4):E45. doi: 10.1542/peds.105.4.e45. PMID 10742366
- [Background] McLaughlin GE, Abitbol CL. Reversal of oliguric tacrolimus nephrotoxicity in children. Nephrol Dial Transplant. 2005 Jul;20(7):1471-5. doi: 10.1093/ndt/gfh785. Epub 2005 Apr 19. PMID 15840666

RESULTS

PARTICIPANT FLOW:
Groups:
- Aminophylline: Patients will receive aminophylline loading dose 5mg/kg prior to transplant and will continue to receive aminophylline 1.8mg/kg Q6h for a total of 20 doses.
  Theophylline drug levels will be monitored daily for 4 days. Target theophylline level is 5-7mcg/ml. Aminophylline dosing will be adjusted in order to achieve desired levels as stated in the study protocol.
Period: Overall Study
Arm/Group | Aminophylline | Control
Started | 23 | 27
Completed | 20 | 25
Not Completed | 3 | 2
Not completed — Physician Decision | 3 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Aminophylline: Patients will receive aminophylline loading dose 5mg/kg prior to transplant and will continue to receive aminophylline 1.8mg/kg Q6h for a total of 20 doses.
  Theophylline drug levels will be monitored daily for 4 days.
  Aminophylline: Aminophylline loading dose 5mg/kg prior to transplant and will continue to receive aminophylline 1.8mg/kg Q6h for a total of 20 doses.
  Theophylline drug levels: Theophylline drug levels will be monitored every morning from all patients for the first 4 days post- transplant.
- Control: Patients will receive placebo infusion of normal saline, pre-transplant, followed by normal saline infusions matched by volume and frequency to treatment arm for a total of 20 doses.
  Drug levels will be monitored daily for 4 days.
  Theophylline drug levels: Theophylline drug levels will be monitored every morning from all patients for the first 4 days post- transplant.
  Placebo: Patients will receive placebo infusion of normal saline, pre-transplant, followed by normal saline infusions matched by volume and frequency to treatment arm for a total of 20 doses.
- Total: Total of all reporting groups
Arm/Group | Aminophylline | Control | Total
Number analyzed (Participants) | 23 | 27 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.28 (4.8) | 11.91 (5.4) | 11.62 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 13 | 15 | 28
Region of Enrollment [Number; unit: participants]
  United States | 23 | 27 | 50

OUTCOME MEASURES:

1. Primary Outcome: Calculated Estimated Glomerular Filtration Rate (eGFR)
Description: The investigators will measure blood creatinine on post-operative day 5 and using the Schwartz equation will calculate estimated glomerular filtration rate (GFR) to determine kidney function.
Time Frame: 5 days
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: ml/min/1.73m2
Arm/Group | Aminophylline | Control
Number analyzed (Participants) | 23 | 27
ml/min/1.73m2 | 67.39 (38.9) | 80.48 (52.1)
Statistical Analysis 1: Comparison: Aminophylline vs Control; Intention to treat analysis; Test type: Superiority — Our calculations showed that by enrolling 50 patients we will be able to detect a 25cc/min absolute difference in eGFR between the two arms with power above 80%, and a two-sided Type I probability error of <0.05; p = 0.32, t-test, 2 sided

2. Secondary Outcome: Urinary NGAL (Neutrophil Gelatinase-associated Lipocalin)/ Creatinine Ratio
Description: urinary NGAL(Neutrophil gelatinase-associated lipocalin) is a biomarker for kidney injury. NGAL levels 12h post-transplant were found to be a marker for development of delayed graft function and need for dialysis post-transplant. NGAL levels are corrected for urine creatinine.
Time Frame: 12 hours post transplant
Population: Participants with available data were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ng/mg
Arm/Group | Aminophylline | Control
Number analyzed (Participants) | 21 | 24
ng/mg | 300.5 [105.5 to 1464.5] | 425.4 [140.3 to 1126.2]
Statistical Analysis 1: Comparison: Aminophylline vs Control; Test type: Superiority — Enrolling 25 patients in each group will allow us to detect a difference of 200ng/mg cr in urinary NGAL levels between the two groups with a power of 80% and a two-sided type I probability error of 0.05; p = 0.95, Kruskal-Wallis

3. Other Pre Specified Outcome: Presence of Fibrosis Measured on Protocol Biopsy
Description: The investigators will use the same cores that are obtained during routine 6 months protocol biopsies to quantify the amount of fibrosis
Time Frame: 6 months
Population: Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Aminophylline | Control
Number analyzed (Participants) | 23 | 26
Participants | 11 | 14
Statistical Analysis 1: Comparison: Aminophylline vs Control; Test type: Superiority; p = 0.67, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Aminophylline | Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/27
Other Adverse Events (participants affected / at risk) | 9/23 | 13/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aminophylline (N=23) | Control (N=27)
Agitation (Nervous system disorders) | 0 | 2
tachycardia at day 1 post transplant (Cardiac disorders) | 7 | 6
tacrolimus toxicity (Injury, poisoning and procedural complications) | 7 | 10
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Rejection (Renal and urinary disorders) | 4 | 6

LIMITATIONS AND CAVEATS:
Small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes